CLINICAL TRIAL: NCT01634854
Title: Randomized Comparison of Vaginal Misoprostol and Intravenous Oxytocin for Labor Induction in Multiparous Women
Brief Title: A Study Comparing Vaginal Misoprostol and Intravenous Oxytocin for Induction of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Angela Wilson-Liverman, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120660
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Induction of Labor in Multiparous Women
MeSH Terms: interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaginal Misoprostol (Active Comparator): Dosage: 25 µg every 4 hours up to a maximum of 4 doses until cervical change is consistent with a diagnosis of active labor Route of administration: Intravaginal
  Interventions: Drug: Vaginal Misoprostol
- Intravenous Oxytocin (Active Comparator): 2 miu per minute increased in increments of 1-2 miu per minute every 30 minutes to establish an effective contraction pattern.
  Route of administration: intravenous
  Interventions: Drug: Intravenous Oxytocin

INTERVENTIONS:
Drug: Vaginal Misoprostol — Dosage: 25 µg every 4 hours up to a maximum of 4 doses until cervical change is consistent with a diagnosis of active labor Route of administration: Intravaginal
  Other Names: Cytotec
  Arms: Vaginal Misoprostol
Drug: Intravenous Oxytocin — Dosage: 2 miu per minute increased in increments of 1-2 miu per minute every 30 minutes to establish an effective contraction pattern.
  Route of administration: intravenous
  Other Names: Pitocin
  Arms: Intravenous Oxytocin

SUMMARY:
This study will compare the effectiveness of vaginal misoprostol (Cytotec) and intravenous oxytocin (Pitocin) in multiparous women who present at term for labor induction.

DETAILED DESCRIPTION:
Both oxytocin and misoprostol have been demonstrated to be safe and effective methods for induction of labor. A direct comparison of efficacy and time to delivery in multiparas has not been specifically investigated. Additionally, the study will look at costs of the two drugs.Oxytocin is administered through an IV so requires more direct patient care time from the Registered Nurse, IV pump, and tubing, whereas misoprostol is a tablet, administered only once, per vagina or orally, every 4 hours. Misoprostol is also very inexpensive comparatively; if equally or more efficacious than oxytocin, this could demonstrate quite a cost and time savings to Vanderbilt University Medical Center and other institutions. Safety of either drug is not in question.

ELIGIBILITY:
Inclusion Criteria:

* Clinical candidate for labor induction utilizing either misoprostol or oxytocin
* Greater than or equal to 18 years of age
* Multiparous
* Singleton gestation;
* Greater than 37 weeks gestation;
* Cephalic presentation

Exclusion Criteria:

* Any clinical contraindication to misoprostol as induction drug
* Age less than 18 years
* Contraindication to vaginal birth
* Nonreassuring fetal heart rate tracing
* Prior uterine surgery
* Active labor
* Active maternal bleeding
* Chorioamnionitis (infection)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Wilson-Liverman, MSN, CNM, Principal Investigator — Vanderbilt University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaudhuri S, Mitra SN, Banerjee PK, Biswas PK, Bhattacharyya S. Comparison of vaginal misoprostol tablets and prostaglandin E2 gel for the induction of labor in premature rupture of membranes at term: a randomized comparative trial. J Obstet Gynaecol Res. 2011 Nov;37(11):1564-71. doi: 10.1111/j.1447-0756.2011.01575.x. Epub 2011 Jun 16. PMID 21676083
- [Background] Olagbuji BN, Ezeanochie MC, Kubeyinje W, Dunsin T, Ande AB. Pregnancy outcome following induction of labor with intravaginal misoprostol for decreased fetal movements at term. J Matern Fetal Neonatal Med. 2011 Oct;24(10):1225-7. doi: 10.3109/14767058.2011.572309. Epub 2011 Apr 20. PMID 21506657
- [Background] Saeed GA, Fakhar S, Nisar N, Alam AY. Misoprostol for term labor induction: a randomized controlled trial. Taiwan J Obstet Gynecol. 2011 Mar;50(1):15-9. doi: 10.1016/j.tjog.2009.08.001. PMID 21482368
- [Background] Shakya R, Shrestha J, Thapa P. Safety and efficacy of misoprostol and dinoprostone as cervical ripening agents. JNMA J Nepal Med Assoc. 2010 Jan-Mar;49(177):33-7. PMID 21180218
- [Background] Hofmeyr GJ, Gulmezoglu AM, Pileggi C. Vaginal misoprostol for cervical ripening and induction of labour. Cochrane Database Syst Rev. 2010 Oct 6;2010(10):CD000941. doi: 10.1002/14651858.CD000941.pub2. PMID 20927722
- [Background] Crane JM, Butler B, Young DC, Hannah ME. Misoprostol compared with prostaglandin E2 for labour induction in women at term with intact membranes and unfavourable cervix: a systematic review. BJOG. 2006 Dec;113(12):1366-76. doi: 10.1111/j.1471-0528.2006.01111.x. PMID 17081181
- [Background] Lin MG, Nuthalapaty FS, Carver AR, Case AS, Ramsey PS. Misoprostol for labor induction in women with term premature rupture of membranes: a meta-analysis. Obstet Gynecol. 2005 Sep;106(3):593-601. doi: 10.1097/01.AOG.0000172425.56840.57. PMID 16135593
- [Background] Li XM, Wan J, Xu CF, Zhang Y, Fang L, Shi ZJ, Li K. Misoprostol in labour induction of term pregnancy: a meta-analysis. Chin Med J (Engl). 2004 Mar;117(3):449-52. PMID 15043790

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Oxytocin: 2 miu per minute increased in increments of 1-2 miu per minute every 30 minutes to establish an effective contraction pattern.
  Route of administration: intravenous
  Intravenous Oxytocin: Dosage: 2 miu per minute increased in increments of 1-2 miu per minute every 30 minutes to establish an effective contraction pattern.
  Route of administration: intravenous
Period: Overall Study
Arm/Group | Vaginal Misoprostol | Intravenous Oxytocin
Started | 64 | 66
Completed | 62 | 59
Not Completed | 2 | 7
Not completed — Cesarean delivery | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaginal Misoprostol | Intravenous Oxytocin | Total
Number analyzed (Participants) | 62 | 59 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 59 | 121
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 59 | 121
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 56 | 55 | 111
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 10 | 26
  White | 43 | 46 | 89
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 59 | 121

OUTCOME MEASURES:

1. Primary Outcome: Time From Induction to Vaginal Delivery
Description: Comparing the time to delivery in multiparas undergoing induction of labor with vaginal misoprostol or intravenous oxytocin.
Time Frame: Time to delivery in minutes from initiation of medication, up to 24 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Vaginal Misoprostol | Intravenous Oxytocin
Number analyzed (Participants) | 62 | 59
minutes | 800 [516 to 1107] | 693 [481 to 884]
Statistical Analysis 1: Comparison: Vaginal Misoprostol vs Intravenous Oxytocin; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Neonatal APGAR Scores
Description: APGAR is a scoring system that evaluates Activity, Pulse, Grimace, Appearance, and Respiration. Each category is given a score of 0-2 points (with 0 being absent and 2 being normal), the points are then combined for a total score that ranges from 0-10. Scores 7 and above are generally normal, 4 to 6 are fairly low, and 2 and below are considered critically low.
Time Frame: At 1 minute and 5 minutes after delivery
Measure: Median (Inter-Quartile Range); unit: number
Arm/Group | Vaginal Misoprostol | Intravenous Oxytocin
Number analyzed (Participants) | 62 | 59
number
  APGAR 1 minute | 8 [8 to 8] | 8 [8 to 8]
  APGAR 5 minute | 9 [9 to 9] | 9 [9 to 9]

3. Secondary Outcome: Neonatal Weight at Delivery
Description: Neonatal Weight
Time Frame: Immediately following delivery
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Vaginal Misoprostol | Intravenous Oxytocin
Number analyzed (Participants) | 62 | 59
grams | 3500 [3082 to 3849] | 3415 [3182 to 3792]

4. Secondary Outcome: Maternal Delivery Outcomes
Description: Maternal delivery outcomes
Time Frame: Through discharge from hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Misoprostol | Intravenous Oxytocin
Number analyzed (Participants) | 62 | 59
Participants
  Epidural | 56 | 48
  Hemorrhage | 2 | 3
  Chorioamnionitis | 2 | 0
  Cesarean delivery | 2 | 7
  Forceps delivery | 4 | 4

5. Secondary Outcome: Maternal Satisfaction With Labor
Time Frame: 6 weeks post-partum
Population: data was not collected
Arm/Group | Vaginal Misoprostol | Intravenous Oxytocin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Excessive Uterine Activity Necessitating Treatment
Description: Number of patients receiving terbutaline during labor for uterine tachysytole
Time Frame: Measured from initiation of medication until delivery time
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Misoprostol | Intravenous Oxytocin
Number analyzed (Participants) | 62 | 59
Participants | 9 | 4

7. Secondary Outcome: NICU Admission and APGAR Less Than 7 at 5 Minutes
Description: NICU admission and APGAR less than 7 at 5 minutes
Time Frame: Through discharge from hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Misoprostol | Intravenous Oxytocin
Number analyzed (Participants) | 62 | 59
Participants
  NICU Admission | 8 | 4
  APGAR less than 7 at 5 min | 0 | 0

ADVERSE EVENTS:
Time Frame: 13 months
Arm/Group | Vaginal Misoprostol | Intravenous Oxytocin
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/59
Other Adverse Events (participants affected / at risk) | 0/62 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes